CLINICAL TRIAL: NCT01602029
Title: Randomized Double Blind Placebo Controlled Study of Ondansetron and Simvastatis Added to Treatment As Usual in Patients with Schizophrenia
Brief Title: Randomized Double Blind Placebo Control Study in Patients with Schizophrenia
Acronym: ROSES
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pakistan Institute of Living and Learning (Other)
Collaborators: Stanley Medical Research Institute (Other); Dow University of Health Sciences (Other); Abbasi Shaheed Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: roses_pill
Record Dates: First submitted 2012-05-17; First posted 2012-05-18 (Estimated); Last update posted 2024-12-10 (Actual); Status verified 2012-05

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Psychosis Not Otherwise Specified; Schizophreniform Disorder
Keywords: Anti inflammatory; Schizophrenia; Simvastatin; Ondansetron
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Ondansetron; Simvastatin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Ondansetron (Active Comparator): ondansetron added to TAU Ondansetron will be administered in 8mg once daily dose
  Interventions: Drug: Ondansetron
- Simvastatin (Active Comparator): Simvastatin added to TAU Simvastatin 20mg taken as once daily dose
  Interventions: Drug: Simvastatin
- Placebo (Placebo Comparator): Placebo added to TAU
  Interventions: Drug: Placebo
- Odansetron Plus Simvastatin (Active Comparator): Ondansetron will be administered in 8mg once daily dose and Simvastatin 20mg taken as once daily dose
  Interventions: Drug: Odansetron plus simvastatin

INTERVENTIONS:
Drug: Ondansetron — ondansetron added to TAU Ondansetron will be administered in 8mg once daily dose
  Arms: Ondansetron
Drug: Simvastatin — Simvastatin added to TAU Simvastatin 20mg taken as once daily dose
  Arms: Simvastatin
Drug: Placebo — Placebo added to TAU
  Arms: Placebo
Drug: Odansetron plus simvastatin — Ondansetron will be administered in 8mg once daily dose and Simvastatin 20mg taken as once daily dose
  Arms: Odansetron Plus Simvastatin

SUMMARY:
Negative symptoms and cognitive deficits are two partially-related features of schizophrenia which have a major negative impact on social function and objective quality of life. Standard drug treatments have little impact on either and arguably no effect on primary negative symptoms. Social dysfunction has major economic consequences in both the developed and developing world. There is evidence that anti-inflammatory treatment may have beneficial effects in patients with schizophrenia.

DETAILED DESCRIPTION:
Negative symptoms and cognitive deficits are two partially-related features of schizophrenia which have a major negative impact on social function and objective quality of life. Evidence indicates that anti-inflammatory treatment may have beneficial effects in schizophrenia. From our preliminary randomised double-blind placebo-controlled clinical trial in Pakistan and Brazil, it is indicated that addition of minocycline (an antibiotic and anti-inflammatory drug) for one year to treatment as usual (TAU) reduced negative symptoms and improved some cognitive measures (Chaudhry et al 2009).

Statins are primarily HMG-CoA reductase inhibitors also anti-inflammatory agents and known to decrease C-reactive protein (CRP). Higher levels of CRP (>0.50 mg/dl) are associated with marked negative symptoms and higher total PANSS scores in patients with schizophrenia. (Fan et al 2007)

Ondansetron, a selective 5-hydroxytryptamine-3 antagonist, is quite commonly used as an antiemetic in cancer patients (Marty et al 1990). There are several small trials suggesting that ondansetron as an adjunct to antipsychotics is effective in improving negative symptoms and memory in patients suffering from schizophrenia (Ahkonzadeh et al 2009, Levkovitz et al 2005 and Zhang et al 2006).

The Primary objective of this study is addition of ondansetron and /or simvastatin to TAU for patients with schizophrenia will result in improvement in negative symptoms

The Secondary objectives include:

* improvement in positive or other symptoms
* social functioning
* cognitive functions
* additive effects of ondansetron and simvastatin

ELIGIBILITY:
Inclusion Criteria

1. Patients aged 18 to 65 years
2. Patients will be recruited both from inpatients and outpatients.
3. Diagnostic and Statistical Manual-IV (DSM-IV TR) diagnosis of schizophrenia, schizoaffective disorder, psychosis not otherwise specified or schizophreniform disorder
4. Competent and willing to give informed consent
5. Stable on medication 4 weeks prior to baseline
6. No planned medication change
7. Able to take oral medication and likely to complete the required evaluations
8. Female participants of child bearing age must be willing to use adequate contraceptives for the duration of the study, and, willing to have a pregnancy test pre treatment and at ten weekly intervals while on study medication,
9. Not planning to relocate in the next 12 months

Exclusion Criteria

1. Relevant ICD 10 organic brain disease or neurological diagnoses (including ECG conduction abnormalities, neurological disorder, or an active seizure)
2. Subjects who will meet the criteria for a DSM-IV TR diagnosis of alcohol or substance abuse (other than for nicotine) within the last month or the criteria for DSM-IV TR alcohol or substance dependence (other than for nicotine) within the last 6 months
3. Any change of psychotropic medications within the previous 4 weeks
4. Pregnant or lactating women and those of reproductive age without adequate contraception

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 303 (Actual)
Dates: Start 2010-08; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Negative symptom severity | 6 months
  Negative symptom severity as defined by negative syndrome subscale score on the Positive and Negative Syndrome Scale

SECONDARY OUTCOMES:
cognitive functioning | 6 months
  1. Full PANSS and positive syndrome subscale score
  2. Clinical Global Impression
  3. Functional outcome

CONTACTS AND LOCATIONS:
Overall Officials: Imran Chaudhry, MD, Principal Investigator — University of Manchester
Locations (3):
- Pakistan (3):
  - Abbasi Shaheed Hospital, Karachi, Sindh
  - Dow university of Health Sciences, Karachi, Sindh
  - Karwan e hayat, Karachi

REFERENCES:
- [Derived] Chaudhry IB, Husain N, Husain MO, Hallak J, Drake R, Kazmi A, Rahman Ru, Hamirani MM, Kiran T, Mehmood N, Stirling J, Dunn G, Deakin B. Ondansetron and simvastatin added to treatment as usual in patients with schizophrenia: study protocol for a randomized controlled trial. Trials. 2013 Apr 17;14:101. doi: 10.1186/1745-6215-14-101. PMID 23782463
- See also: Website of Pakistan Institute of Learning & Living — http://pill.org.pk